CLINICAL TRIAL: NCT01836172
Title: Multicenter, Randomized, Double Blind, Placebo-controlled, Phase II Clinical Trial to Evaluate the Safety and Efficacy of YJP-14 Capsules for the Treatment of Endothelial Dysfunction in Patients With Diabetes Mellitus
Brief Title: YJP-14 Capsules for the Treatment of Endothelial Dysfunction in Patients With Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Han Wha Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HW2012-YJP002
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Complication
Keywords: The treatment of diabetic complication
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo t.i.d. (Placebo Comparator): Placebo t.i.d.
  Interventions: Drug: YJP-14
- YJP-14 25 mg t.i.d. (Placebo Comparator): YJP-14 25 mg t.i.d. YJP-14 is a 50% ethanolic extract of Lindera obtusiloba stems.
  Interventions: Drug: YJP-14
- YJP-14 50 mg t.i.d. (Placebo Comparator): YJP-14 50 mg t.i.d. YJP-14 is a 50% ethanolic extract of Lindera obtusiloba stems.
  Interventions: Drug: YJP-14
- YJP-14 100 mg t.i.d. (Placebo Comparator): YJP-14 is a 50% ethanolic extract of Lindera obtusiloba stems. YJP-14 100 mg t.i.d.
  Interventions: Drug: YJP-14

INTERVENTIONS:
Drug: YJP-14 — An 50% ethanolic extract of Lindera obtusiloba stems
  Other Names: An 50% ethanolic extract of Lindera obtusiloba stems

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of YJP-14 capsules for the treatment of endothelial dysfunction in patients with diabetes mellitus.

DETAILED DESCRIPTION:
The primary purpose of this study is to demonstrate superior effect of YJP-14 three doses, 25, 50 and 100 mg t.i.d on endothelial dysfunction in diabetes mellitus indicated as mean change difference of flow-mediated dilation (FMD), compared to placebo group after treatment of 12 weeks.

The secondary purposes of this study are divided into three as follows;

* Clinically significant effect of YJP-14 three doses, 25, 50 and 100 mg t.i.d on endothelial dysfunction in diabetes mellitus indicated as mean change difference of FMD, compared to placebo group after treatment of 8 weeks.
* Clinically significant effect of YJP-14 three doses, 25, 50 and 100 mg t.i.d on insulin resistance in diabetes mellitus indicated as mean change difference of Homeostasis Model Assessment-Insulin Resistance (HOMA-IR), compared to placebo group after treatment of 4, 8 and 12 weeks.
* Clinically significant effect of YJP-14 three doses, 25, 50 and 100 mg t.i.d on mean change difference of blood pressure in diabetes mellitus, compared to placebo group after treatment of 4, 8 and 12 weeks.

The exploratory purposes of this study are divided into two as follows;

* Clinically significant effect of YJP-14 three doses, 25, 50 and 100 mg t.i.d on blood glucose level in diabetes mellitus indicated as mean change difference of HbA1c, compared to placebo group after treatment of 12 weeks.
* Clinically significant effect of YJP-14 three doses, 25, 50 and 100 mg t.i.d on vascular stiffness in diabetes mellitus indicated as mean change difference of blood lipids (LDL, HDL and TG), compared to placebo group after treatment of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Adult-onset DM (defined as fasting glucose greater than 125 mg/dl or by ongoing treatment with an oral hypoglycemic agent), Endothelial dysfunction: FMD below 6.7%, LDL cholesterol level less than 140 mg/dl, Patients agreed to Informed Consent Form

Exclusion Criteria: (Key exclusion criteria) Uncontrolled arterial hypertension (above 139/90 mmHg) or hypotension (below 80/50 mmHg), Severe diabetic complication: diabetic nephropathy, diabetic neuropathy, diabetic retinopathy, diabetic vascular complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Flow-mediated dilation (FMD) | 12 weeks

SECONDARY OUTCOMES:
Flow-mediated dilation (FMD) Homeostasis Model Assessment-Insulin Resistance (HOMA-IR) Systolic and Diastolic Blood Pressure | 8 weeks
Homeostasis model assessment-insulin resistance (HOMA-IR) | 4, 8, 12 weeks
Systolic and Diastolic Blood Pressure | 4, 8, 12 weeks

OTHER OUTCOMES:
HbA1c Serum lipids (LDL, HDL and TG) | 12 weeks
Serum Lipids (LDL, HDL and TG) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Hee Oh, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Internal medicine, Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Lee JO, Oak MH, Jung SH, Park DH, Auger C, Kim KR, Lee SW, Schini-Kerth VB. An ethanolic extract of Lindera obtusiloba stems causes NO-mediated endothelium-dependent relaxations in rat aortic rings and prevents angiotensin II-induced hypertension and endothelial dysfunction in rats. Naunyn Schmiedebergs Arch Pharmacol. 2011 Jun;383(6):635-45. doi: 10.1007/s00210-011-0643-9. Epub 2011 May 2. PMID 21533989
- [Background] Lee JO, Auger C, Park DH, Kang M, Oak MH, Kim KR, Schini-Kerth VB. An ethanolic extract of Lindera obtusiloba stems, YJP-14, improves endothelial dysfunction, metabolic parameters and physical performance in diabetic db/db mice. PLoS One. 2013 Jun 3;8(6):e65227. doi: 10.1371/journal.pone.0065227. Print 2013. PMID 23755196